CLINICAL TRIAL: NCT06671327
Title: Preemptive Analgesia Of Dexmedetomidine Reduces Per-operation Pain After Noncardiac Surgery
Brief Title: Preemptive Analgesia Of Dexmedetomidine Reduces Per-operation Pain
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: China International Neuroscience Institution (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Health Services Research
Other Study IDs: CINI-AD-2024-0112
Record Dates: First submitted 2024-07-25; First posted 2024-11-04 (Actual); Last update posted 2025-04-09 (Actual); Status verified 2025-03

CONDITIONS: Pain Management; Noncardiac Surgery
MeSH Terms: conditions — Agnosia | interventions — Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Dexmedetomidine group (Experimental): The DEX group was continuously pumped at 1.5 μg /(kg·h) for 15 minutes before induction, and after induction continue infusion 15min.
  Interventions: Drug: Preemptive Dexmedetomidine injection
- Placebo group (Placebo Comparator): the Placebo group was infused with equal amounts of 0.9% Sodium Chloride
  Interventions: Drug: Sodium Chloride 0.9% Inj

INTERVENTIONS:
Drug: Preemptive Dexmedetomidine injection — The DEX group was continuously pumped at 1.5 μg /(kg·h) for 15 minutes before induction, and after induction continue infusion 15min.
  Other Names: Preemptive Dex
  Arms: Dexmedetomidine group
Drug: Sodium Chloride 0.9% Inj — The Placebo group was infused with equal amounts of isochronous normal saline.
  Other Names: Preemptive Sodium Chloride 0.9%
  Arms: Placebo group

SUMMARY:
Background:Preemptive analgesia is the initiation of analgesic regimen before the onset of nociceptive stimulation, preventing the amplification of pain due to peripheral and central sensitization and thereby reducing subsequent pain. Preemptive analgesia of dexmedetomidine (DEX) in the epidural and subarachnoid space can effectively prevent the central sensitization, and significantly reduce the phantom limb pain, residual pain after one year of lower limb amputation.

Objective: To investigate the per-operative effects of DEX preemptive analgesia.

Method:The patients scheduled noncardiac surgery undergoing general anesthesia were selected and divided into DEX group and Placebo group randmized. The DEX group was continuously pumped at 1.5 μg /(kg·h) for 15 minutes before induction, and 15min after induction. The Placebo group was infused with equal amounts of normal saline.The Coprimary efficacy outcome was a composite of analgesia effect, one is the Compliance Rate of IOC2 target in intra-operation, another is the the rate of none-to-slight post-operative pain assessed with the p-NRS≦3 at 12 hours after surgery [Pain numeric rating scale was assessed with the (Numeric Rating Scale, p-NRS)].

DETAILED DESCRIPTION:
Background:Preemptive analgesia is the initiation of analgesic regimen before the onset of nociceptive stimulation, preventing the amplification of pain due to peripheral and central sensitization and thereby reducing subsequent pain. Preemptive analgesia of DEX in the epidural and subarachnoid space can effectively prevent the central sensitization, and significantly reduce the phantom limb pain, residual pain after one year of lower limb amputation.

Objective: To investigate the per-operative effects of DEX preemptive analgesia.

ELIGIBILITY:
Inclusion Criteria:

* 18 years to 85 years old,
* body mass index (BMI,calculated as weight in kilograms divided by height in meters squared): 18.5~35.
* ASA (American Society of Anesthesiologists) Grade I- III;
* Scheduled for non-cardiac surgery undergoing general anesthesia
* expected duration of operation 0.5~3 h.

Exclusion Criteria:

* disagreed to participate;
* body mass index (BMI) of greater 35
* American Society of Anesthesiologists (ASA) classification 4 or above;
* previous severe central nervous systemheart, liver, kidney or and lung dysfunction ;
* diagnosed neuropsychological disorders, that is, schizophrenia, epilepsy, Parkinson's disease, myasthenia gravis，Alzheimer's disease and other autonomic disorders of patients affecting EEG outcomes;
* comatose, dementia, or language barrier which impeded communication and assessment;
* history of neurosurgical procedures;
* Systolic blood pressure continuously lower than 85mmHg or higher than 180mmHg; heart rate continuously lower than 45 times / min; sever arrhythmia need intervation and implantable pacemaker.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 208 (Estimated)
Dates: Start 2025-04-03 (Estimated); Primary Completion 2025-06-23 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
The coprimary efficacy outcome | During the whole operation
  The rate of intro-operative IOC2 target reachment
The coprimary efficacy outcome | post-operative 24 hours
  The rate of none-to-slight post-operative pain, assessed with the (Numeric Rating Scale)p-NRS< =3 at 24h post-opertively.
The primary safety outcome | During 48 h post-operation
  Adverse events and safety outcomes within during 48 h post-operation: hypotension, Hypertension,Bradycardia,Tachycardia,Respiratory depression,Pulse oxygen desaturation and the number of patients which need intervention.

SECONDARY OUTCOMES:
SBP | During the whole operation
  systolic blood pressure(intraoperative hemodynamics)
DBP | During the whole operation
  dystolic blood pressure(intraoperative hemodynamics)
MAP | During the whole operation
  mean arterial pressure(intraoperative hemodynamics)
HR | During the whole operation
  Heart rate (intraoperative hemodynamics)
Bispectral index | During the whole operation
  Bispectral index
EMG | During the whole operation
  Electromyogram Index
pNRS at Hour 0, Hour 24, Hour 48, and the Day 7 postoperatively | post-operation p-NRS until 7 days(inculde Hour 0, Hour 24, Hour 48, and the Day 7 timepoints)
  Record and compared the pNRS at Hour 0, Hour 24, Hour 48, and the Day 7 postoperatively. (The p-NRS was an 11-point scale with 0 indicating no pain and 10 equaled worst pain).
mPONV | Postoperative immediately and until 12 hours post-operatively
  modified postoperative nausea vomiting (mPONV) score at postoperative immediately (0 hour)and 24 hours post-operatively.
  Modified PONV Scoring Criteria:
  0 points: No nausea or vomiting.
  1. point: Nausea present, no vomiting.
  2. points: Nausea with one vomiting episode. Additional points: +1 per additional vomiting episode (e.g., 4 vomiting episodes = 5 points).
The accumulation of analgesia consumption | Hour 24, Hour 48, and the Day 7 after surgery
  The accumulation of analgesia consumption was used to describe oxycodone accumulation (oral administration of oxycodone 5 mg for each complaint of pain) at Hour 24, Hour 48, and the Day 7 after surgery.
Dizziness | Hour 0, Hour 24 and the Hour 48 post-operatively
  Dizziness at Hour 0, Hour 24 and the Hour 48 post-operatively
Agitation | immediately afer surgery(Hour 0 post-operation)
  Agitation immediately afer surgery(Hour 0 post-operation)
The rate of exhaust | until 24hours post-operation
  The rate of exhaust at first 24hours post-operation
Extubation time | after operation immediately
  Extubation time

CONTACTS AND LOCATIONS:
Locations (1):
- Xuanwu hospital, Beijing, Beijing Municipality, China